CLINICAL TRIAL: NCT00428402
Title: Using Focus Groups to Assess the Impact of Environmental Health Science Programs for K-12 Educational Community
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0125
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Education; 4th-8th Grade Student; MIDAS Project; Focus Group Discussion; Bastrop

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Focus Group: Participant is a 4th-8th grade student in select schools from Bastrop Independent School District (BISD).
  Interventions: Behavioral: Focus Group Discussion

INTERVENTIONS:
Behavioral: Focus Group Discussion — Focus groups meeting for up to 1 hour during the regular school day.

SUMMARY:
The MIDAS Project (Models of Implementation and Dissemination of Environmental Health and Science Across Subjects) Assessment Objectives:

* Determine whether students are aware of the MIDAS Project.
* Identify strengths and weaknesses of MIDAS Project components including: integrated environmental health and science (EHS) curricula, field experiences, seminars and student projects.
* Assess career interests and intended courses of study at the college level.

DETAILED DESCRIPTION:
You are being asked to give your child permission to take part in a focus group to talk about what he or she has learned over the past year. Your child's school and other schools in the area have been working with a program called the Models of Implementation and Dissemination of Environmental Health and Science Across Subjects (MIDAS) Project. The MIDAS Project was developed by The University of Texas M.D. Anderson Cancer Center, Smithville, TX.

Purpose:

Students will be asked to share about the topics that they learned about over the past year, including their field trip experiences. Participation in the focus group is strictly voluntary, and your child may or may not choose to take part. This focus group will not be graded, and your child's name will not be recorded with his or her responses. If your child chooses not to participate in this focus group, he or she will not be penalized in any way.

ELIGIBILITY:
Inclusion Criteria:

* Students must be in one of the identified classes in one of the participating grades from one of the participating schools.
* Students must return a completed and signed parental consent form.
* Students must be present at school on the day that the focus groups are conducted.

Exclusion Criteria:

* Students whose parents did not complete the consent form, and/or students who do not wish to participate can opt out of the focus groups without any penalty.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participant is a 4th-8th grade student in select schools from Bastrop Independent School District (BISD).
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2007-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Outputs From Focus Groups (Qualitative Narrative) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Robin Fuchs-Young, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org